CLINICAL TRIAL: NCT01286272
Title: A Randomized Phase II Trial of Ofatumumab and Bendamustine vs. Ofatumumab, Bortezomib (NSC # 681239) and Bendamustine in Patients With Untreated Follicular Lymphoma
Brief Title: Ofatumumab and Bendamustine Hydrochloride With or Without Bortezomib in Treating Patients With Untreated Follicular Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02625; NCI-2011-02625 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CALGB-50904; CDR0000694298; CALGB-50904 (Other: Alliance for Clinical Trials in Oncology); CALGB-50904 (Other: CTEP); U10CA031946 (NIH); U10CA180821 (NIH)
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Results first posted 2019-01-10 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Ann Arbor Stage III Grade 1 Follicular Lymphoma; Ann Arbor Stage III Grade 2 Follicular Lymphoma; Ann Arbor Stage III Grade 3 Follicular Lymphoma; Ann Arbor Stage IV Grade 1 Follicular Lymphoma; Ann Arbor Stage IV Grade 2 Follicular Lymphoma; Ann Arbor Stage IV Grade 3 Follicular Lymphoma; Grade 3a Follicular Lymphoma
MeSH Terms: interventions — Bendamustine Hydrochloride; Bortezomib; Fluorodeoxyglucose F18; ofatumumab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (ofatumumab, bendamustine hydrochloride) (Experimental): INDUCTION: Patients receive ofatumumab IV over 2-8 hours on day 1 and bendamustine hydrochloride IV over 30-60 minutes on days 1 and 2. Treatment repeats every 35 days for up to 6 courses. Patients without disease progression continue on to maintenance therapy.
  MAINTENANCE: Beginning 8 weeks after the start of induction course 6, patients receive ofatumumab IV over 2-8 hours on day 1. Treatment repeats every 56 days for up to 4 courses.
  Interventions: Drug: Bendamustine Hydrochloride; Radiation: Fludeoxyglucose F-18; Other: Laboratory Biomarker Analysis; Biological: Ofatumumab; Procedure: Positron Emission Tomography with Radiolabeled Targeting Agent
- Arm B (ofatumumab, bendamustine hydrochloride, bortezomib) (Experimental): INDUCTION: Patients receive ofatumumab IV over 2-8 hours on day 1, bendamustine hydrochloride IV over 30-60 minutes on days 1 and 2, and bortezomib IV over 3-5 seconds or SC on days 1, 8, 15, and 22. Treatment repeats every 35 days for up to 6 courses. Patients without disease progression continue on to maintenance therapy.
  MAINTENANCE: Beginning 8 weeks after the start of induction course 6, patients receive ofatumumab IV over 2-8 hours on day 1 and bortezomib IV over 3-5 seconds or SC on days 1, 8, 15, and 22. Treatment repeats every 56 days for up to 4 courses.
  Interventions: Drug: Bendamustine Hydrochloride; Drug: Bortezomib; Radiation: Fludeoxyglucose F-18; Other: Laboratory Biomarker Analysis; Biological: Ofatumumab; Procedure: Positron Emission Tomography with Radiolabeled Targeting Agent

INTERVENTIONS:
Drug: Bendamustine Hydrochloride — Given IV
  Other Names: Belrapzo; Bendamustin Hydrochloride; Bendeka; CEP 18083; CEP-18083; CEP18083; Cytostasan Hydrochloride; Levact; Ribomustin; SyB L-0501; Treakisym; Treanda; VIVIMUSTA
Drug: Bortezomib — Given IV or SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; LDP-341; LDP341; MLN 341; MLN-341; MLN341; PS 341; PS-341; PS341; Velcade
  Arms: Arm B (ofatumumab, bendamustine hydrochloride, bortezomib)
Radiation: Fludeoxyglucose F-18 — Undergo FDG-PET
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Ofatumumab — Given IV
  Other Names: Arzerra; GSK1841157; HuMax-CD20; HuMax-CD20, 2F2; Kesimpta
Procedure: Positron Emission Tomography with Radiolabeled Targeting Agent — Undergo FDG-PET
  Other Names: Positron Emission Tomography with Radiolabeled Targeting Agents

SUMMARY:
This randomized phase II trial studies how well ofatumumab and bendamustine hydrochloride with or without bortezomib works in treating patients with untreated follicular non-Hodgkin lymphoma. Monoclonal antibodies, such as ofatumumab, may block cancer growth in different ways by targeting certain cells. Drugs used in chemotherapy, such as bendamustine hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Bortezomib may also stop the growth of cancer cells by blocking blood flow to the tumor. It is not yet known whether ofatumumab and bendamustine hydrochloride are more effective with bortezomib in treating patients with follicular non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the complete response (CR) rate in newly diagnosed, untreated follicular lymphoma patients receiving 6 cycles of ofatumumab-bendamustine (bendamustine hydrochloride) (ARM A) and 6 cycles of ofatumumab, bortezomib, and bendamustine (ARM B) using International Harmonization Project Response Criteria.

SECONDARY OBJECTIVES:

I. To determine progression-free survival (PFS) of patients with untreated follicular lymphoma after 6 cycles of ofatumumab-bendamustine (ARM A) followed by maintenance ofatumumab and after 6 cycles of ofatumumab, bortezomib, and bendamustine followed by maintenance ofatumumab and bortezomib (ARM B).

II. To determine the toxicity profile of ofatumumab and bendamustine and ofatumumab, bortezomib, and bendamustine in patients with untreated high-risk follicular lymphoma.

III. To determine if changes in both qualitative and semi-quantitative fludeoxyglucose (FDG)-positron-emission tomography (PET) findings at baseline, after cycle 2 (day 32-35), and at end of therapy (6-8 weeks after the last cycle of induction chemotherapy but prior to maintenance therapy) with ofatumumab-bendamustine and ofatumumab, bortezomib, and bendamustine correlate with response and PFS in patients with high-risk follicular lymphoma.

IV. To assess if a combinatorial approach using both qualitative and semi-quantitative changes in FDG-PET and computed tomography (CT) or magnetic resonance imaging (MRI) studies at baseline, after cycle 2 (day 32-35), and at end of therapy (6-8 weeks after the last cycle of induction chemotherapy prior to maintenance therapy) would result in a higher predictive value for response and PFS in patients with high-risk follicular lymphoma.

V. To correlate all molecular parameters with FDG-PET parameters in determination of response and PFS.

VI. To correlate pre-treatment single nucleotide polymorphisms with response and PFS following ofatumumab-bendamustine and ofatumumab, bortezomib, and bendamustine therapy in patients with untreated high-risk follicular lymphoma.

VII. To correlate cluster of differentiation (CD)-68, B-cell chronic lymphocytic leukemia (CLL)/lymphoma (bcl)-2, marker of proliferation Ki-67 (Ki-67), forkhead box P3 (FOXP3), activated cytotoxic T-cells, lymphoma-associated macrophages (LAM), melanoma associated antigen (mutated) 1 (MUM1), CD10, nuclear v-rel avian reticuloendotheliosis viral oncogene homolog A (p65) and v-rel avian reticuloendotheliosis viral oncogene homolog C (cREL) subunits of nuclear factor of kappa light polypeptide gene enhancer in B-cells (NFkB), and selected genetic translocations by fluorescent in situ hybridization (FISH) analysis (such as Bcl-2 and Bcl-6) with response and PFS in patients receiving initial therapy for high-risk follicular lymphoma.

VIII. To determine whether immune gene signatures previously identified as prognostic factors in follicular lymphoma can be applied to paraffin-embedded tissues in ofatumumab and bendamustine or ofatumumab, bendamustine, and bortezomib treated patients; evaluate micro-ribonucleic acid (RNA) signatures associated with these gene signatures and outcome.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A:

INDUCTION: Patients receive ofatumumab intravenously (IV) over 2-8 hours on day 1 and bendamustine hydrochloride IV over 30-60 minutes on days 1 and 2. Treatment repeats every 35 days for up to 6 courses. Patients without disease progression continue on to maintenance therapy.

MAINTENANCE: Beginning 8 weeks after the start of induction course 6, patients receive ofatumumab IV over 2-8 hours on day 1. Treatment repeats every 56 days for up to 4 courses.

ARM B:

INDUCTION: Patients receive ofatumumab IV over 2-8 hours on day 1, bendamustine hydrochloride IV over 30-60 minutes on days 1 and 2, and bortezomib IV over 3-5 seconds or subcutaneously (SC) on days 1, 8, 15, and 22. Treatment repeats every 35 days for up to 6 courses. Patients without disease progression continue on to maintenance therapy.

MAINTENANCE: Beginning 8 weeks after the start of induction course 6, patients receive ofatumumab IV over 2-8 hours on day 1 and bortezomib IV over 3-5 seconds or SC on days 1, 8, 15, and 22. Treatment repeats every 56 days for up to 4 courses.

After completion of study treatment, patients are followed up every 4 months for 2 years and then every 6 months for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed follicular non-Hodgkin lymphoma, World Health Organization (WHO) classification grade 1, 2, or 3a (> 15 centroblasts per high-power field with centrocytes present)

  * Bone marrow biopsies as the sole means of diagnosis are not acceptable, but they may be submitted in conjunction with nodal biopsies
  * Fine-needle aspirates are not acceptable
  * Failure to submit pathology within 60 days of patient registration will be considered a major protocol violation
* Patients must have at least one of the following indicators of poor risk disease:

  * >= 3 risk factors by the Follicular Lymphoma International Prognostic Index, or 2 risk factors by the Follicular Lymphoma International Prognostic Index and at least one bulky mass or lymph node > 6 cm in size
  * Follicular Lymphoma International Prognostic Index (FLIPI score):

    * Age > 60 years
    * Involvement of > 4 nodal sites
    * Stage III-IV disease
    * Hemoglobin < 12.0 g/dL
    * Lactate dehydrogenase (LDH) > upper limit of normal (ULN)

      * 0-1 of the above risk factors: low risk
      * 2 risk factors: intermediate risk
      * >= 3 risk factors: poor risk
* No prior cytotoxic chemotherapy, radiotherapy, immunotherapy, or radioimmunotherapy
* No corticosteroids are permitted, except for maintenance therapy for a non-malignant disease or to prevent treatment-related ofatumumab reactions (maintenance therapy dose must not exceed 20 mg/day prednisone or equivalent)
* Measurable disease must be present either on physical examination or imaging studies; non-measurable disease alone is not acceptable; any tumor mass > 1 cm is acceptable; lesions that are considered non-measurable include the following:

  * Bone lesions
  * Leptomeningeal disease
  * Ascites
  * Pleural/pericardial effusion
  * Inflammatory breast disease
  * Lymphangitis cutis/pulmonis
  * Bone marrow involvement (involvement by non-Hodgkin lymphoma should be noted)
* Patients must have no known central nervous system (CNS) involvement by lymphoma
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must be non-pregnant and non-nursing; pregnant or nursing patients may not be enrolled; women of childbearing potential must have a negative serum or urine pregnancy test within 14 days prior to registration; in addition, women and men of childbearing potential must commit to use an effective form of contraception throughout their participation in this study; appropriate methods of birth control include abstinence, oral contraceptives, implantable hormonal contraceptives (Norplant), or double barrier method (diaphragm plus condom)
* Patients with human immunodeficiency virus (HIV) infection are eligible; patients with HIV infection must meet the following: no evidence of co-infection with hepatitis B or C; CD4+ count > 400/ul; no evidence of resistant strains of HIV; on anti-HIV therapy with an HIV viral load < 50 copies HIV RNA/mL; no history of acquired immunodeficiency syndrome (AIDS)-defining conditions; no zidovudine or stavudine are allowed owing to overlapping toxicity with chemotherapy
* Patients must have no evidence of active hepatitis B or C infection (i.e., no positive serology for anti-hepatitis B core [HBc] or anti-hepatitis C virus [HCV] antibodies); hepatitis B virus (HBV) seropositive patients (hepatitis B surface antigen [HBsAg] +) are eligible if HBV deoxyribonucleic acid (DNA) is undetectable at baseline and they are closely monitored for evidence of active HBV infection by HBV DNA testing at each treatment cycle; after completing treatment, HBsAg + patients must be monitored by HBV DNA testing every 2 months for 6 months post-treatment, while continuing lamivudine
* Granulocytes >= 1,000/uL
* Platelet count >= 75,000/uL
* Creatinine =< 2.0 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limits of normal (ULN)
* Bilirubin =< 2 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2011-04-28 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2025-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristie A Blum, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (96):
- United States (96):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Saint Helena Hospital, St. Helena, California
  - Middlesex Hospital, Middletown, Connecticut
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Randolph Hospital, Asheboro, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Altru Cancer Center, Grand Forks, North Dakota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia

REFERENCES:
- [Derived] Rutherford SC, Yin J, Pederson L, Perez Burbano G, LaPlant B, Shadman M, Li H, LeBlanc ML, Kenkre VP, Hong F, Blum KA, Dockter T, Martin P, Jung SH, Grant B, Rosenbaum C, Ujjani C, Barr PM, Unger JM, Cheson BD, Bartlett NL, Kahl B, Friedberg JW, Mandrekar SJ, Leonard JP. Relevance of Bone Marrow Biopsies for Response Assessment in US National Cancer Institute National Clinical Trials Network Follicular Lymphoma Clinical Trials. J Clin Oncol. 2023 Jan 10;41(2):336-342. doi: 10.1200/JCO.21.02301. Epub 2022 Jul 5. PMID 35787017
- [Derived] Blum KA, Polley MY, Jung SH, Dockter TJ, Anderson S, Hsi ED, Wagner-Johnston N, Christian B, Atkins J, Cheson BD, Leonard JP, Bartlett NL. Randomized trial of ofatumumab and bendamustine versus ofatumumab, bendamustine, and bortezomib in previously untreated patients with high-risk follicular lymphoma: CALGB 50904 (Alliance). Cancer. 2019 Oct 1;125(19):3378-3389. doi: 10.1002/cncr.32289. Epub 2019 Jun 7. PMID 31174236

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One hundred thirty five patients registered to this trial. However, 3 patients cancelled prior to receiving any study treatment and were excluded from all analyses.
Groups:
- Arm A (Ofatumumab, Bendamustine Hydrochloride): INDUCTION: Patients receive:> 300 mg ofatumumab IV over 2-8 hours on day 1, cycle1 and 1000 mg ofatumumab IV on day 1, cycle 2-6 and 90 mg/m2 bendamustine hydrochloride IV over 30-60 minutes on days 1 and 2. Treatment repeats every 35 days for up to 6 courses. Patients without disease progression continue on to maintenance therapy. >
  > MAINTENANCE: Beginning 8 weeks after the start of induction course 6, patients receive 1000 mg ofatumumab IV over 2-8 hours on day 1. Treatment repeats every 56 days for up to 4 courses.
- Arm B (Ofatumumab, Bendamustine Hydrochloride, Bortezomib): INDUCTION: Patients receive 300 mg ofatumumab IV over 2-8 hours on day 1, cycle1 and 1000 mg ofatumumab IV on day 1, cycle 2-6 and 90 mg/m2 bendamustine hydrochloride IV over 30-60 minutes on days 1 and 2, and 1.6 mg/m2 bortezomib IV over 3-5 seconds or SC on days 1, 8, 15, and 22. Treatment repeats every 35 days for up to 6 courses. Patients without disease progression continue on to maintenance therapy. >
  > MAINTENANCE: Beginning 8 weeks after the start of induction course 6, patients receive 1000 mg ofatumumab IV over 2-8 hours on day 1 and 1.6 mg/m2 bortezomib IV over 3-5 seconds or SC on days 1, 8, 15, and 22. Treatment repeats every 56 days for up to 4 courses.
Period: Overall Study
Arm/Group | Arm A (Ofatumumab, Bendamustine Hydrochloride) | Arm B (Ofatumumab, Bendamustine Hydrochloride, Bortezomib)
Started | 67 | 65
Completed | 66 | 62
Not Completed | 1 | 3
Not completed — Ineligible after beginning treatment | 1 | 3

BASELINE CHARACTERISTICS:
Population: All patients that were eligible for endpoint analysis were included in the baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Ofatumumab, Bendamustine Hydrochloride) | Arm B (Ofatumumab, Bendamustine Hydrochloride, Bortezomib) | Total
Number analyzed (Participants) | 66 | 62 | 128
Age, Continuous [Median (Full Range); unit: years] | 61 [25 to 87] | 61.5 [31 to 81] | 61 [25 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 32 | 60
  Male | 38 | 30 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 62 | 56 | 118
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 54 | 58 | 112
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 4 | 16
Region of Enrollment [Number; unit: participants]
  United States | 66 | 62 | 128

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: A complete response was defined using International Harmonization Project Response Criteria as the complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. If the bone marrow was involved by lymphoma before treatment, the infiltrate must have cleared on repeat bone marrow biopsy.
  The complete response (CR) rate was calculated in newly diagnosed untreated follicular lymphoma patients receiving 6 cycles of ofatumumab-bendamustine (ARM A) and 6 cycles of ofatumumab, bortezomib, and bendamustine (ARM B).
  The complete response rate was calculated as the number of patients with a complete response divided by the number of patients eligible for evaluation.
Time Frame: From date of randomization until patient stops treatment for any reason, up to 484 days post-randomization
Population: All patients that were eligible for response assessment were included in this analysis.
Measure: Number; unit: proportion of patients
Groups:
- Arm A (Ofatumumab, Bendamustine Hydrochloride): INDUCTION: Patients receive:
  300 mg ofatumumab IV over 2-8 hours on day 1, cycle1 and 1000 mg ofatumumab IV on day 1, cycle 2-6 and 90 mg/m2 bendamustine hydrochloride IV over 30-60 minutes on days 1 and 2. Treatment repeats every 35 days for up to 6 courses. Patients without disease progression continue on to maintenance therapy.
  MAINTENANCE: Beginning 8 weeks after the start of induction course 6, patients receive 1000 mg ofatumumab IV over 2-8 hours on day 1. Treatment repeats every 56 days for up to 4 courses.
- Arm B (Ofatumumab, Bendamustine Hydrochloride, Bortezomib): INDUCTION: Patients receive 300 mg ofatumumab IV over 2-8 hours on day 1, cycle1 and 1000 mg ofatumumab IV on day 1, cycle 2-6 and 90 mg/m2 bendamustine hydrochloride IV over 30-60 minutes on days 1 and 2, and 1.6 mg/m2 bortezomib IV over 3-5 seconds or SC on days 1, 8, 15, and 22. Treatment repeats every 35 days for up to 6 courses. Patients without disease progression continue on to maintenance therapy.
  MAINTENANCE: Beginning 8 weeks after the start of induction course 6, patients receive 1000 mg ofatumumab IV over 2-8 hours on day 1 and 1.6 mg/m2 bortezomib IV over 3-5 seconds or SC on days 1, 8, 15, and 22. Treatment repeats every 56 days for up to 4 courses.
Arm/Group | Arm A (Ofatumumab, Bendamustine Hydrochloride) | Arm B (Ofatumumab, Bendamustine Hydrochloride, Bortezomib)
Number analyzed (Participants) | 66 | 62
proportion of patients | .621 | .597

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. PFS rates (percentages) at 1, 2, ,3 and 4 years are defined as the percentage of patients who are alive and progression-free at the respective time points. The p-values of the log-rank test will be calculated to compare PFS between the two arms.
Time Frame: Up to 4 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A (Ofatumumab, Bendamustine Hydrochloride) | Arm B (Ofatumumab, Bendamustine Hydrochloride, Bortezomib)
Number analyzed (Participants) | 66 | 62
percentage of patients
  PFS at 1 year | 93.8 [88.2 to 99.9] | 84.8 [76.2 to 94.5]
  PFS at 2 years | 80.3 [70.8 to 91.0] | 75.6 [65.2 to 87.7]
  PFS at 3 years | 65.9 [53.9 to 80.7] | 67.1 [55.5 to 81.0]
  PFS at 4 years | 57.3 [43.2 to 75.9] | 64.7 [52.8 to 79.2]
Statistical Analysis 1: Comparison: Arm A (Ofatumumab, Bendamustine Hydrochloride) vs Arm B (Ofatumumab, Bendamustine Hydrochloride, Bortezomib); Test type: Superiority; p = 0.8457, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.51 to 1.74]

3. Secondary Outcome: The Number of Patients Who Experienced Grade 3+ Hematologic and Non-hematologic Adverse Events at Least Possibly Related to Treatment
Description: The number of patients who experienced grade 3+ hematologic and non-hematologic adverse events at least possibly related to treatment assessed according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0
Time Frame: From date of randomization until patient stops treatment for any reason, up to 484 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Ofatumumab, Bendamustine Hydrochloride) | Arm B (Ofatumumab, Bendamustine Hydrochloride, Bortezomib)
Number analyzed (Participants) | 66 | 62
Participants
  Hematologic | 45 | 41
  Non-Hematologic | 17 | 33

4. Other Pre Specified Outcome: Pre-treatment Single Nucleotide Polymorphisms (SNP)
Description: The PFS will be compared among the three genotype groups of each SNP using the log-rank tests. A maxtype test will be used by taking the maximum value of the log-rank tests under dominant, recessive, and proportional hazard model. The critical value (or p-value) of the max test will be obtained by a permutation method. No multiple testing adjustment may be applied because of the small sample size.
Time Frame: Up to 10 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Immunohistochemical (IHC) Markers
Description: The IHC markers will be correlated with response (using the two-sample t-test) and PFS (using the Cox regression method) data. No multiple testing adjustment will be applied because of the small sample size.
Time Frame: Up to 10 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Predictive Value of Fludeoxyglucose-positron-emission Tomography
Description: The ratio will be correlated with response (using the two-sample t-test) and PFS (using the Cox regression method) data.
Time Frame: Up to 36-38 weeks (6-8 weeks after course 6, day 1 after last course of induction chemotherapy)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected systematically after each cycle, up to 10 cycles. Cycles 1-6 were up to 35 days and cycles 7-10 were up to 56 days.
Arm/Group | Arm A (Ofatumumab, Bendamustine Hydrochloride) | Arm B (Ofatumumab, Bendamustine Hydrochloride, Bortezomib)
All-Cause Mortality (participants affected / at risk) | 1/67 | 4/65
Serious Adverse Events (participants affected / at risk) | 1/67 | 4/65
Other Adverse Events (participants affected / at risk) | 67/67 | 65/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Ofatumumab, Bendamustine Hydrochloride) (N=67) | Arm B (Ofatumumab, Bendamustine Hydrochloride, Bortezomib) (N=65)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Ofatumumab, Bendamustine Hydrochloride) (N=67) | Arm B (Ofatumumab, Bendamustine Hydrochloride, Bortezomib) (N=65)
Anemia (Blood and lymphatic system disorders) | 30 (141) | 40 (149)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 3 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (4)
Chest pain - cardiac (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 4 (5)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (8)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 4 (5)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (6) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (4) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 4 (16) | 10 (27)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 4 (6)
Dry eye (Eye disorders) | 2 (2) | 6 (12)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 1 (2)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 4 (5)
Eye pain (Eye disorders) | 0 (0) | 2 (3)
Flashing lights (Eye disorders) | 0 (0) | 1 (1)
Floaters (Eye disorders) | 1 (6) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 2 (4)
Watering eyes (Eye disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 21 (37) | 13 (27)
Anal fistula (Gastrointestinal disorders) | 1 (3) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 2 (2) | 2 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 25 (71) | 34 (130)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 22 (61) | 39 (116)
Dry mouth (Gastrointestinal disorders) | 2 (13) | 6 (28)
Dyspepsia (Gastrointestinal disorders) | 15 (38) | 11 (28)
Dysphagia (Gastrointestinal disorders) | 4 (7) | 1 (2)
Esophageal pain (Gastrointestinal disorders) | 3 (6) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 2 (3)
Flatulence (Gastrointestinal disorders) | 4 (8) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (6)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 (16) | 4 (5)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (9) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 11 (12) | 9 (11)
Nausea (Gastrointestinal disorders) | 39 (125) | 55 (192)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 4 (11) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 2 (3) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 12 (20) | 33 (57)
Chills (General disorders) | 8 (9) | 18 (32)
Edema face (General disorders) | 1 (1) | 2 (2)
Edema limbs (General disorders) | 11 (16) | 9 (19)
Edema trunk (General disorders) | 0 (0) | 1 (1)
Facial pain (General disorders) | 1 (2) | 1 (1)
Fatigue (General disorders) | 49 (241) | 46 (207)
Fever (General disorders) | 11 (16) | 24 (35)
Flu like symptoms (General disorders) | 2 (2) | 4 (4)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 3 (3)
Infusion related reaction (General disorders) | 15 (19) | 13 (16)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 2 (2)
Irritability (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 1 (6) | 3 (4)
Malaise (General disorders) | 4 (4) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (5) | 3 (3)
Pain (General disorders) | 10 (19) | 17 (42)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Allergic reaction (Immune system disorders) | 27 (35) | 30 (37)
Anaphylaxis (Immune system disorders) | 1 (1) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 10 (11) | 6 (8)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 1 (5) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Cecal infection (Infections and infestations) | 1 (2) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 4 (11)
Infections and infestations - Other, specify (Infections and infestations) | 6 (8) | 8 (11)
Lung infection (Infections and infestations) | 3 (4) | 4 (4)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 2 (5) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 7 (9) | 2 (3)
Skin infection (Infections and infestations) | 4 (6) | 7 (9)
Small intestine infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 12 (26) | 7 (16)
Urinary tract infection (Infections and infestations) | 7 (8) | 5 (6)
Bruising (Injury, poisoning and procedural complications) | 4 (8) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (9)
Alanine aminotransferase increased (Investigations) | 20 (75) | 10 (23)
Alkaline phosphatase increased (Investigations) | 5 (11) | 6 (11)
Aspartate aminotransferase increased (Investigations) | 24 (61) | 14 (52)
Blood bilirubin increased (Investigations) | 8 (15) | 2 (2)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 5 (15)
Cardiac troponin I increased (Investigations) | 1 (4) | 0 (0)
Cholesterol high (Investigations) | 1 (5) | 3 (7)
Creatinine increased (Investigations) | 12 (32) | 14 (42)
Ejection fraction decreased (Investigations) | 2 (5) | 0 (0)
GGT increased (Investigations) | 0 (0) | 1 (1)
INR increased (Investigations) | 3 (7) | 2 (2)
Investigations - Other, specify (Investigations) | 3 (9) | 3 (7)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 48 (284) | 44 (218)
Lymphocyte count increased (Investigations) | 1 (1) | 3 (14)
Neutrophil count decreased (Investigations) | 40 (130) | 35 (119)
Platelet count decreased (Investigations) | 32 (140) | 35 (136)
Weight gain (Investigations) | 5 (11) | 4 (10)
Weight loss (Investigations) | 7 (15) | 8 (19)
White blood cell decreased (Investigations) | 37 (198) | 43 (183)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 16 (42) | 18 (54)
Dehydration (Metabolism and nutrition disorders) | 6 (8) | 9 (16)
Hypercalcemia (Metabolism and nutrition disorders) | 5 (11) | 7 (16)
Hyperglycemia (Metabolism and nutrition disorders) | 28 (135) | 25 (78)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (9) | 4 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 2 (3) | 2 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 4 (8) | 6 (16)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (9) | 11 (16)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (20) | 11 (23)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (6) | 5 (11)
Hypokalemia (Metabolism and nutrition disorders) | 9 (20) | 16 (22)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (11) | 6 (11)
Hyponatremia (Metabolism and nutrition disorders) | 7 (14) | 12 (14)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (9) | 3 (5)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 4 (17) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (45) | 10 (20)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (22) | 15 (42)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (14) | 6 (15)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8 (26) | 7 (18)
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3 (14) | 2 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (28) | 9 (22)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (12) | 4 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (43) | 8 (24)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 0 (0)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (6) | 0 (0)
Concentration impairment (Nervous system disorders) | 1 (8) | 0 (0)
Dizziness (Nervous system disorders) | 15 (24) | 17 (36)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 11 (30) | 6 (19)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (3)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 14 (42) | 18 (43)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (2)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 3 (3) | 4 (5)
Movements involuntary (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (3) | 1 (3)
Neuralgia (Nervous system disorders) | 1 (2) | 4 (12)
Olfactory nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (2) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 7 (10)
Peripheral sensory neuropathy (Nervous system disorders) | 16 (62) | 36 (146)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Sinus pain (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (2) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 3 (5)
Tremor (Nervous system disorders) | 2 (11) | 1 (1)
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 13 (47) | 16 (28)
Confusion (Psychiatric disorders) | 2 (2) | 3 (5)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 7 (13) | 4 (10)
Insomnia (Psychiatric disorders) | 17 (50) | 13 (50)
Libido decreased (Psychiatric disorders) | 1 (8) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (3) | 3 (4)
Proteinuria (Renal and urinary disorders) | 2 (3) | 5 (6)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 2 (3)
Urinary frequency (Renal and urinary disorders) | 3 (7) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 2 (9) | 2 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (2)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 6 (11) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (47) | 18 (41)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (38) | 16 (46)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (7)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 7 (12)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (7) | 2 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (18) | 6 (13)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (3) | 3 (12)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (21) | 12 (17)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 21 (48) | 25 (51)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 6 (9) | 5 (6)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 2 (2)
Hot flashes (Vascular disorders) | 4 (12) | 6 (16)
Hypertension (Vascular disorders) | 18 (79) | 13 (42)
Hypotension (Vascular disorders) | 5 (9) | 12 (17)
Phlebitis (Vascular disorders) | 1 (2) | 2 (4)
Superficial thrombophlebitis (Vascular disorders) | 1 (1) | 1 (2)
Thromboembolic event (Vascular disorders) | 3 (4) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/72/NCT01286272/Prot_SAP_000.pdf